CLINICAL TRIAL: NCT03689517
Title: Placebo Modulation of Orthodontic Pain: a Single-blind Functional MRI Study
Brief Title: Placebo Modulation of Orthodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meiya Gao, Principal Investigator, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2014-048
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo arm (Experimental): Orthodontic pain was introduced by placement of orthodontic elastic separators to the mesial and distal sides of the right mandibular first molar. Participants took placebos (pills made by starch) that were told to be an effective analgesic
  Interventions: Other: placebo; Device: orthodontic elastic separators
- sham arm (Sham Comparator): Orthodontic pain was introduced by placement of orthodontic elastic separators to the mesial and distal sides of the right mandibular first molar. But participants do not take placebos
  Interventions: Device: orthodontic elastic separators

INTERVENTIONS:
Other: placebo — participants took placebos (pills made by starch) that were told to be an effective analgesic.
  Arms: placebo arm
Device: orthodontic elastic separators — Orthodontic pain was introduced by placement of orthodontic elastic separators to the mesial and distal sides of the right mandibular first molar.

SUMMARY:
How placebo modulates orthodontic pain remains largely unknown. The present study aimed to investigate the placebo modulation of brain activity associated with orthodontic pain using fMRI.

DETAILED DESCRIPTION:
How placebo modulates orthodontic pain remains largely unknown. The present study aimed to investigate the placebo modulation of brain activity associated with orthodontic pain using fMRI. 23 voluneers were recruited in a longitudinal fMRI experiment. At both the baseline and the one-month follow-up, orthodontic separators were placed between right lower molars 24 hours before MRI scans. At baseline, the subjects were scanned without placebo while all subjects took placebos half an hour before the scan at follow-up. Scans include a bite/non-bite task fMRI and a followed resting state fMRI. A generalized linear model was used to identify pain-regulating network from task fMRI, and functional connectivity analysis of pain related brain regions was performed to study the possible modulation of placebo on connectivity of pain-regulating networks using resting-state fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Female, 20-25 years old;
* Right handed;
* Understand the Visual Analog Scale;
* No history of serious illness, surgery, psychiatric disorders or neurological;
* No history of drug or alcohol abuse;
* No Maxillofacial diseases, agomphiasis, caries, metal filling material or crown;
* Individual normal occlusion with no orthodontic treatment history.

Exclusion Criteria:

* claustrophobic or experienced obvious adverse reactions including fear, nausea, vomiting
* discomfort during the scan process or during menstruation.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
fMRI data change during MRI scan | Day 1
  The fMRI data were collected with a Siemens 3.0T MRI system at West China Hospital. Scans include a bite/non-bite task fMRI and a followed resting state fMRI. Through MRI data we can investigate the modulation of brain activity associated with orthodontic pain using fMRI.

SECONDARY OUTCOMES:
The chronological changes of anxiety level | Day 1
  Secondary outcomes concerning chronological changes of anxiety were assessed before and after orthodontic treatments through state-trait anxiety inventory (ST-AI). A higher score indicates higher anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Wenli Lai, Prof, Study Director — West China hospital of stomatology

IPD SHARING:
Plan to Share IPD: No